CLINICAL TRIAL: NCT00629057
Title: An Open-Label, Phase I Dose Escalation Trial of MVA-BN®-PRO in Men With Androgen-Insensitive Prostate Cancer
Brief Title: A Safety Trial of MVA-BN®-PRO in Men With Androgen-Insensitive Prostate Cancer
Acronym: BNIT-PR-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNIT-PR-001
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2011-06

CONDITIONS: Androgen-insensitive Prostate Cancer
Keywords: androgen-insensitive, non-metastatic, prostate, cancer
MeSH Terms: conditions — Neoplasms | interventions — MVA-BN-PRO vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Lowest dose level
  Interventions: Biological: MVA-BN-PRO
- 2 (Experimental): Middle level dose
  Interventions: Biological: MVA-BN-PRO
- 3 (Experimental): Highest dose level
  Interventions: Biological: MVA-BN-PRO

INTERVENTIONS:
Biological: MVA-BN-PRO — 1x10e8 TCID50 q 4 wks x 6
  Arms: 1
Biological: MVA-BN-PRO — 2 x 10e8 TCID50 q 4 wks x 6
  Arms: 2
Biological: MVA-BN-PRO — 4 x 10e8 TCID50 q 4 wks x 6
  Arms: 3

SUMMARY:
BNIT-PR-001 is an open-label, multi-center, Phase I dosing evaluation trial of MVA-BN®-PRO in men with androgen-insensitive prostate cancer. Patients will have PSA recurrence after being treated with androgen suppression therapy or complete androgen blockade.

The trial will consist of a treatment with up to 6 vaccinations with MVA-BN®-PRO at monthly intervals, followed by a 1-year follow-up phase. A vaccination may be 1, 2, or 4 injections of study vaccine.

The study is designed to examine safety as well as the effect of three different doses on immune response.

DETAILED DESCRIPTION:
MVA-BN®-PRO is a candidate prostate cancer immunotherapy product comprised of a highly attenuated non-replicating vaccinia virus, MVA-BN®, engineered to encode prostate specific antigen (PSA) and prostate acid phosphatase (PAP) proteins. The MVA-BN®-based vaccine provides innate and adaptive immune activating factors, and vaccination by this strategy will be evaluated for its capacity to help override self and tumor tolerance mechanisms.

Previous work has shown PSA and PAP antigens to be immunogenic in humans when presented with immune stimulatory components. Multiple clinical studies have demonstrated promising activity of PSA-targeted vaccinia-based immunotherapy. Additionally, PAP-based cellular therapy immunization approaches, have shown promise in Phase III clinical trials and provided for enhanced survival. The strategy undertaken by BNIT is to combine both antigens in the MVA-BN® vector to enhance the immunogenic effect and to help mitigate development of tumor resistance.

This trial examines three vaccination regimens of MVA-BN®-PRO:

Vaccine is provided at (0.5cc/dose/1x10e8 TCID50)

* Cohort 1: 1 sc injection every 4 weeks x 3; retreated once at the same dose and schedule.
* Cohort 2: 2 sc injections every 4 weeks x 3; retreated once at the same dose and schedule.
* Cohort 3: 4 sc injections every 4 weeks x 3; retreated once at the same dose and schedule.

These dose regimens are based on the current dose of MVA-BN® (1x10e8 TCID50 by sc injection) under development as a prophylactic vaccine for the prevention of smallpox, and on related clinical studies of MVA-nef-based vaccines (5x10e8 TCID50) for induction of heterologous immunity.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men, 18 - 75 years of age
* Documented prostate cancer with a rising PSA post androgen suppression or blockade therapy
* Chemotherapy naïve
* ECOG Performance Score of 0,1, or 2
* Life expectancy ≥ 1 year
* No significant cardiac, bone marrow, hepatic, or renal dysfunction; or coagulopathy (defined as no AE ≥ Grade 3 according to NCI CTCAE v 3.0). Patients with a known history of a CLINICALLY NON-SIGNIFICANT laboratory parameter may be eligible for inclusion provided an exemption is granted by the study Medical Monitor prior to enrollment.
* A negative virology screen for HIV, hepatitis B surface antigen, and hepatitis C

Exclusion Criteria:

* Metastatic disease
* Congestive heart failure (NYHA Class III or IV), unstable angina, or cardiovascular disease such as stroke or myocardial infarction (current or within the past 6 months)
* History of prior malignancies other than prostate cancer within the past 5 years, excluding basal or squamous cell carcinoma of the skin
* Known allergy to eggs, egg products, or aminoglycoside antibiotics, e.g., gentamicin or tobramycin
* Chronic administration (defined as 5 or more days of consecutive use) of systemic corticosteroids within 14 days of the first planned dose of MVA-BN®-PRO. Use of inhaled steroids, nasal sprays, eye drops and topical creams for small body areas is allowed.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement hormones are not excluded.
* Prior solid organ or hematopoietic allogenic transplant(s)
* Receipt of an investigational agent within 28 days of the first planned dose of MVA-BN®-PRO
* Prior "vaccine" therapy for prostate cancer at any time
* Vaccination: Live (attenuated) vaccine (e.g., FluMist®). Vaccination with a live vaccine within 28 days of the first planned dose of MVA-BN®-PRO, or plans to receive a live vaccine within 28 days after the last dose of MVA-BN®-PRO is not allowed
* Vaccination: Killed (inactivated) vaccine (e.g., PneumoVax®). Vaccination with a killed vaccine within 14 days of the first planned dose of MVA-BN®-PRO, or plans to receive a killed vaccine within 14 days after the last dose of MVA-BN®-PRO is not allowed.
* Radiation therapy within 28 days of the first planned dose of MVA-BN®-PRO or plans for radiation therapy during treatment or re-treatment. Prior to initiating palliative radiation during the (re)treatment phase of the study, the Sponsor's medical monitor or designee must be notified.
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints
* Study personnel

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple injection regimens of MVA-BN®-PRO for the treatment of androgen-insensitive prostate cancer. | Continuous

SECONDARY OUTCOMES:
To evaluate the ability of MVA-BN®-PRO to generate humoral and cellular immune responses to prostate antigens, and to define an optimal dose for future studies. | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, Study Director — Bavarian Nordic
Locations (7):
- United States (7):
  - Urology Centers of Alabama, Homewood, Alabama
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Presbyterian Hospital Center for Cancer Research, Charlotte, North Carolina
  - Urology Associates, Nashville, Tennessee
  - Urology Clinics of North Texas, PA, Dallas, Texas
  - Urology Associates of South Texas, McAllen, Texas